CLINICAL TRIAL: NCT02233517
Title: Group Cognitive Behavioral Therapy for Anger and Aggression in Veterans With PTSD
Brief Title: Group CBT for Aggression in Veterans
Acronym: CBT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1298-W; 1IK2RX001298-01A2 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-09-08 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Aggression; Anger; Posttraumatic Stress Disorder
Keywords: Veterans; Cognitive-Behavioral Therapy; Aggression; Anger; Posttraumatic Stress Disorder; Combat Disorders
MeSH Terms: conditions — Aggression; Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive-Behavioral Therapy for Anger and Aggression in Combat Veterans with PTSD (CBT-A) is a 12-week manualized group treatment protocol that is grounded in up-to-date research, and that specifically addresses the Energy and Drive Functions, Attention Functions, Emotion Functions, and Thought Functions that are hypothesized to underlie the limitations to Activities and Participation associated with PTSD-related anger and aggression. Each session lasts 90 minutes. The first session orients participants to the structure and philosophy of the program, provides a historical overview of PTSD, and introduces the concept of the "survival mode" of functioning (Chemtob et al., 1997). The remaining 11 sessions follow a standard format: 1) practice relaxation training (15-20 minutes); 2) review homework, introduce new material, and engage in group activities focused on implementing new skills and behaviors (70-80 minutes); and 3) review problems or concerns of group members.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Present Centered Therapy (Active Comparator): Present Centered Therapy (PCT) is an active, manualized treatment comparison condition for psychotherapy trials. PCT is designed to control for nonspecific factors of therapy such as contact with a trained therapist, rationale for treatment, and instillation of expectancy for therapeutic gains. The therapeutic approach was drawn from Yalom's group therapy model, which utilizes interpersonal process, supportive techniques, identification of response options, encouragement of adaptive reactions, and focus on the "here-and-now". Previous large-scale randomized clinical trials of Veterans with PTSD have found reduced PTSD symptoms in the PCT comparison condition (Schnurr et al., 2003), and a survey of practice patterns within the VA suggests that similar present-focused approaches are routinely employed by VA mental health providers (Rosen et al., 2004). Consistent with recommendations in the PCT manual, training will emphasize the approach rather than specific interventions.
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy provides patients with the skills to 1) identify and challenge maladaptive cognitions that are contributing to self-destructive behaviors; and 2) implement techniques such as relaxation training, communication skills, and relaxation training to address physiological and environmental barriers to effective functioning.
  Arms: Cognitive Behavioral Therapy
Behavioral: Present Centered Therapy — Present Centered Therapy utilizes interpersonal process, supportive techniques, identification of response options, encouragement of adaptive reactions, and focus on the "here-and-now" to support patients in their efforts to improve functioning.
  Arms: Present Centered Therapy

SUMMARY:
Posttraumatic stress disorder (PTSD) robustly predicts anger and aggression, and U.S. Iraq/Afghanistan-era combat Veterans report that treatment for anger and aggression is among their top priorities. PTSD-related anger and aggression are associated with profound functional impairments, yet to date there are no empirically-supported treatments for Veterans with PTSD and aggression. Effective group treatment programs could improve functioning and facilitate community reintegration for these Veterans. Given that anger impedes progress in treatment of PTSD symptoms, group anger treatment could also improve Veterans' capacity to benefit from individually-administered empirically-supported therapy for PTSD such as prolonged exposure or cognitive processing therapy.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) robustly predicts anger and aggression (Olatunji, Ciesielski, & Tolin, 2010), and U.S. Iraq/Afghanistan-era Veterans report that controlling anger and aggressive urges are primary readjustment concerns (Sayer et al, 2010). Trauma-related anger and aggression are associated with functional impairments that significantly limit community reintegration (Rodriguez, Holowka, & Marx, 2012) and that may persist for decades (Koenen et al, 2003). As more troops return from multiple deployments to Iraq and Afghanistan, there is an urgent and growing need for the development and testing of psychosocial treatment for anger and aggression in combat Veterans with PTSD. VA clinicians are doing their best to be responsive to Veteran's needs by offering anger management treatment to Veterans: A survey of clinical practices within the VA found that 35-65% of VA PTSD specialists report providing anger management to their patients (Rosen et al., 2004). Yet to date only one randomized clinical trial (RCT), published in 1997, has investigated the efficacy of treatment of anger and aggression in Veterans with PTSD (Chemtob et al., 1997).

A recent review noted that most researchers who have examined the effects of anger management interventions have not done so as part of a systematic program of research (DiGiuseppe and Tafrate, 2003). The proposed CDA-2 application outlines Training and Mentoring Plans that will provide the applicant with the foundation to establish a career systematically developing, testing, and refining treatments for PTSD-related anger and aggression in Veterans. The following specific Training Goals have been formulated: 1) To acquire the advanced skills in the development and evaluation of clinical interventions necessary to begin an independent research career within the VA; 2) To develop greater expertise in delivery of behavioral interventions to improve functional outcomes and community reintegration in Veterans with PTSD, anger problems, and aggression; 3) To acquire expertise in the development and evaluation of treatment innovations to help Veterans generalize treatment gains beyond the therapy setting; 4) To increase understanding of rehabilitation theory and methods in treatment practices and research; and 5) To achieve critical professional development milestones, including submission of a Merit Review proposal based on the pilot data generated from the CDA-2 project.

The Research Plan proposes a pilot feasibility trial for an RCT of Cognitive-Behavioral Therapy for Anger and Aggression in Combat Veterans with PTSD (CBT-A). CBT-A is a 12-week manualized group treatment protocol that has been designed to address the specific needs of combat Veterans whose PTSD-related anger and aggression interfere with effective community reintegration. The group was implemented with 4 male Vietnam Veterans with severe combat-related PTSD who were referred for anger management treatment, and preliminary data were promising. The active comparison treatment for the pilot RCT will be group Present-Centered Therapy (PCT), a manualized treatment for PTSD that controls for treatment time, social support, and instillation of hope. The proposed research project will address the following Specific Aims: Aim 1: Characterize the differential effects of group CBT-A and group PCT on anger, aggression, and anger/aggression-related limitations to psychosocial functioning and community reintegration in combat Veterans with PTSD; and Aim 2: Evaluate study feasibility and treatment delivery procedures of an RCT comparing CBT-A to a PCT comparison condition. The results generated will guide the design of a full RCT to be funded by the end of the CDA-2 funding period. The research, training, and mentoring plans outlined here will provide the foundation for the PI's independent research career developing a systematic program of research in the treatment of anger and aggression among combat Veterans with PTSD. The availability of empirically-supported anger treatment would benefit the many Veterans with PTSD who return from combat reporting problems with anger and aggression.

ELIGIBILITY:
Inclusion Criteria:

A Veteran will meet criteria for inclusion if he/she meets all of the following criteria:

* Current PTSD based on the CAPS;
* served in combat (regardless of era or country of combat service);
* can speak and write fluent conversational English;
* at least 18 years of age;
* report problems with irritability, anger, or aggression within the past month. Problems with anger and aggression will be defined via the "rule of 4": Inclusion in the study will require a CAPS-V score > 2 on item 15 (E1), "irritable or angry and showed it in your behavior" item within the past month.

Exclusion Criteria:

A Veteran will be excluded from participation if he/she:

* is expected to be unstable on his/her medication regimen during the study;
* currently meets criteria for Bipolar I Disorder or a primary psychotic disorder as determined by the Structured Clinical Interview for the DSM (most current version available) (SCID);
* is receiving (or plan to) other anger-management psychotherapy during the course of the study;
* will be undergoing empirically supported psychotherapy for PTSD during the treatment component of the study;
* meets criteria for substance dependence (other than nicotine) within the past month as determined by the SCID; or
* is determined to have moderate or severe impairment related to traumatic brain injury as measured by the Brief Traumatic Brain Injury Screen and consultation with the Veteran's provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Van Voorhees, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dennis PA, Dennis NM, Van Voorhees EE, Calhoun PS, Dennis MF, Beckham JC. Moral transgression during the Vietnam War: a path analysis of the psychological impact of veterans' involvement in wartime atrocities. Anxiety Stress Coping. 2017 Mar;30(2):188-201. doi: 10.1080/10615806.2016.1230669. Epub 2016 Sep 19. PMID 27580161
- [Background] Van Voorhees EE, Dennis PA, Neal LC, Hicks TA, Calhoun PS, Beckham JC, Elbogen EB. Posttraumatic Stress Disorder, Hostile Cognitions, and Aggression in Iraq/Afghanistan Era Veterans. Psychiatry. 2016 Spring;79(1):70-84. doi: 10.1080/00332747.2015.1123593. PMID 27187514
- [Background] Van Voorhees EE, Dennis PA, Elbogen EB, Clancy CP, Hertzberg MA, Beckham JC, Calhoun PS. Personality assessment inventory internalizing and externalizing structure in veterans with posttraumatic stress disorder: associations with aggression. Aggress Behav. 2014 Nov-Dec;40(6):582-92. doi: 10.1002/ab.21554. Epub 2014 Aug 16. PMID 25131806
- [Background] Ulmer CS, Van Voorhees E, Germain AE, Voils CI, Beckham JC; VA Mid-Atlantic Mental Illness Research Education and Clinical Center Registry Workgroup. A Comparison of Sleep Difficulties among Iraq/Afghanistan Theater Veterans with and without Mental Health Diagnoses. J Clin Sleep Med. 2015 Sep 15;11(9):995-1005. doi: 10.5664/jcsm.5012. PMID 26094928
- [Background] Van Voorhees EE, Beckham JC. Advancements in treating intimate partner violence in veterans. J Clin Psychiatry. 2015 Jun;76(6):e826-7. doi: 10.4088/JCP.14com09556. No abstract available. PMID 26132696
- [Background] Tye S, Van Voorhees E, Hu C, Lineberry T. Preclinical perspectives on posttraumatic stress disorder criteria in DSM-5. Harv Rev Psychiatry. 2015 Jan-Feb;23(1):51-8. doi: 10.1097/HRP.0000000000000035. PMID 25563569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were excluded after enrollment: 13 did not meet inclusion criteria; 17 declined to participate or were lost to contact.
Groups:
- Cognitive Behavioral Therapy: Cognitive-Behavioral Therapy for Anger and Aggression in Combat Veterans with PTSD (CBT-A) is a 12-week manualized group treatment protocol Each session lasts 90 minutes.The first session orients participants to the program, provides an overview of PTSD, and introduces the concept of the "survival mode" of functioning. The remaining 11 sessions follow a standard format: 1) practice relaxation training (15-20 minutes); 2) review homework, introduce new material, and engage in group activities focused on implementing new skills and behaviors (70-80 minutes); and 3) review problems or concerns of group members. Cognitive Behavioral Therapy: CBT-A provides patients with the skills to 1) identify and challenge maladaptive cognitions that are contributing to self-destructive behaviors; and 2) implement techniques such as relaxation training, communication skills, and relaxation training to address physiological and environmental barriers to effective functioning.
- Present Centered Therapy: Present Centered Therapy (PCT) is an active, manualized treatment comparison condition for psychotherapy trials. PCT is designed to control for nonspecific factors of therapy such as contact with a trained therapist, rationale for treatment, and instillation of expectancy for therapeutic gains. The therapeutic approach was drawn from Yalom's group therapy model, which utilizes interpersonal process, supportive techniques, identification of response options, encouragement of adaptive reactions, and focus on the "here-and-now". Consistent with recommendations in the PCT manual, training will emphasize the approach rather than specific interventions.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Started | 19 | 17
Completed | 12 | 13
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Therapy: Cognitive-Behavioral Therapy for Anger and Aggression in Combat Veterans with PTSD (CBT-A) is a 12-week manualized group treatment protocol. Each session lasts 90 minutes. The first session orients participants to the structure and philosophy of the program, provides a historical overview of PTSD, and introduces the concept of the "survival mode" of functioning. The remaining 11 sessions follow a standard format: 1) practice relaxation training (15-20 minutes); 2) review homework, introduce new material, and engage in group activities focused on implementing new skills and behaviors (70-80 minutes); and 3) review problems or concerns of group members. CBT-A provides patients with the skills to 1) identify and challenge maladaptive cognitions that are contributing to self-destructive behaviors; and 2) implement techniques such as relaxation training, communication skills, and relaxation training to address physiological and environmental barriers to effective functioning.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.7) | 52.6 (12.3) | 51.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 7 | 7 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Scores on the Conflicts Tactics Scale (CTS) From Baseline to Post-treatment, 3 Month and 6 Month Follow-up.
Description: Physically aggressive behaviors including throwing something at someone, pushing, grabbing, shoving, slapping, kicking, biting, hitting, beating up, threatening with a gun or knife, or using a gun or knife on someone. Scale range 0 (never) to 6 (more than 20 times) over past 30 days.
Time Frame: pre-treatment (baseline), post-treatment (12 weeks), 3 months post-treatment (48 weeks), and 6 months post-treatment (84 weeks)
Population: Last observation carried forward analyses used; 36 participants assigned to groups. Data screening found one participant's data (male, CBT arm) were not valid; 35 participants' data analyzed. One participant (male, PCT arm) contacted, confirmed that 3 month data was invalid; data for this subject, this time point, this measure not used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Present Centered Therapy: Present Centered Therapy (PCT) is an active, manualized treatment comparison condition for psychotherapy trials. PCT is designed to control for nonspecific factors of therapy such as contact with a trained therapist, rationale for treatment, and instillation of expectancy for therapeutic gains. The therapeutic approach was drawn from Yalom's group therapy model, which utilizes interpersonal process, supportive techniques, identification of response options, encouragement of adaptive reactions, and focus on the "here-and-now". Previous large-scale randomized clinical trials of Veterans with PTSD have found reduced PTSD symptoms in the PCT comparison condition (Schnurr et al., 2003), and similar present-focused approaches are routinely employed by VA mental health providers (Rosen et al., 2004). Consistent with recommendations in the PCT manual, training will emphasize the approach rather than specific interventions.
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 0.50 (0.99) | 1.24 (4.13)
  post-treatment | 0.22 (0.73) | 1.06 (4.12)
  3-month follow-up: number analyzed (Participants) | 18 | 16
  3-month follow-up | 0.61 (1.50) | 1.19 (4.23)
  6-month follow-up | 0.94 (2.04) | 1.18 (4.11)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = -0.10, Standard Error of Mean 0.51 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p < 0.44, Mixed Models Analysis; Slope = 0.23, Standard Error of Mean 0.52 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.33, Mixed Models Analysis; Slope = 0.50, Standard Error of Mean 0.51 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

2. Primary Outcome: Change in Mean Scores on the Dimensions of Anger Reactions Scale (DAR) Over 16 Time Points: Baseline, 12 Treatment Sessions, Post-treatment, 3-month and 6-month Follow-up
Description: The DAR is a 7-item scale measuring the frequency, duration, and behavioral response to anger, and anger-related functional impairment on social relationships, health, and work. The scale will be administered weekly to provide information about the pattern of change in anger- and aggression-related cognitions over the course of the group. Scores range from 0 to 56, with higher scores reflecting greater impairment.
Time Frame: pre-treatment (baseline), weekly treatment sessions, post-treatment (12 weeks), 3 months post-treatment (48 weeks), and 6 months post-treatment (84 weeks)
Population: Last observation carried forward analyses used; 36 participants assigned to groups. Data screening found one participant's data (male, CBT arm) were not valid; 35 participants' data analyzed. Data for baseline session incomplete/unscorable for one participant (female, CBT arm); her data not included in outcome means table, so n for CBT arm is 17.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 19 | 17
units on a scale
  baseline: number analyzed (Participants) | 17 | 17
  baseline | 40.2 (12.6) | 41.2 (10.4)
  post-treatment: number analyzed (Participants) | 17 | 17
  post-treatment | 34.6 (14.2) | 36.8 (14.6)
  3 month follow-up: number analyzed (Participants) | 17 | 17
  3 month follow-up | 35.8 (13.2) | 38.2 (13.9)
  6 month follow-up: number analyzed (Participants) | 17 | 17
  6 month follow-up | 35.5 (13.4) | 36.1 (12.7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Multilevel model of therapy type (1=CBT, 2=PCT), gender, and time on DAR scores, using data from baseline, 12 sessions, post-treatment, 3-month and 6-month follow up; Test type: Superiority — Estimation parameter is interaction of session by therapy, or estimate of difference in mean between CBT and PCT per time point. Positive value is less decrease over time in CBT arm (greater decrease in anger over time in PCT); p = 0.26, Mixed Models Analysis; Mean Difference (Net) = 0.11, Standard Error of Mean 0.10

3. Primary Outcome: Change in Mean Scores on the Novaco Anger Scale (NAS) From Baseline to Post-treatment, 3-month Follow-up, and 6-month Follow-up.
Description: The NAS is a measure anger and coping that indexes four aspects of the experience of anger: Cognitive, Arousal, Behavior, and Anger Regulation. The T-score for the total NAS is used as the outcome, with a range of 0 to 100. Higher scores reflect greater impairment.
Time Frame: as for outcome 1
Population: The NAS was not used with the first cohort of CBT, so the total N for this measure is 28. Last observation carried forward used to address missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 11 | 17
units on a scale
  baseline | 74.2 (4.6) | 75.9 (3.1)
  post-treatment | 74.3 (5.0) | 76.1 (3.5)
  3 month follow-up | 74.8 (3.3) | 76.3 (3.0)
  6 month follow-up | 74.7 (2.6) | 76.1 (3.4)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.90, Mixed Models Analysis; Mean Difference (Net) = -0.14, Standard Error of Mean 1.16 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.85, Mixed Models Analysis; Mean Difference (Net) = 0.22, Standard Error of Mean 1.16 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.79, Mixed Models Analysis; Mean Difference (Net) = 0.31, Standard Error of Mean 1.16 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

4. Secondary Outcome: Change in Mean Scores on the Community Reintegration of Service Members Computer Adaptive Test From Baseline to Post-treatment.
Description: The computer-adaptive version of the CRIS was developed specifically to assess the ICF domain of Participation in Veterans. The Perceived Limitations to Participation subscale assesses Veterans' perceived limitations in participation, and includes items such as "I felt that I easily lost control of my feelings". The Extent of Participation subscale assesses how often Veterans experience a challenge in participation, and includes items such as "How often did you get together with friends?" The Satisfaction with Participation subscale assesses Veterans' level of satisfaction with participation, and includes items such as "How satisfied were you with your daily accomplishments?" Each of the scales has a range of 0-100, with higher scores reflecting better functioning.
Time Frame: pre-treatment (baseline), post-treatment (12 weeks)
Population: Last observation carried forward analyses used. Three participants did not have baseline measures, so were not included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 17 | 16
units on a scale
  Baseline, Perceived Limitations | 41.1 (3.5) | 41.0 (4.6)
  Post-treatment, Perceived Limitations | 40.7 (3.2) | 41.1 (5.9)
  Baseline, Extent of Participation | 38.4 (6.3) | 37.9 (7.9)
  Post-treatment, Extent of Participation | 37.7 (5.8) | 39.5 (8.5)
  Baseline, Satisfacation | 41.4 (3.6) | 40.7 (3.4)
  Post-treatment, Satisfaction | 41.6 (3.7) | 41.6 (4.4)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; This is the comparison of change in means for cognitive-behavioral vs. present-centered therapy from baseline to post-treatment for the Extent of Participation scale; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Net) = -2.3, 95% CI 2-sided [-4.5 to -.002], Standard Deviation 3.2
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; This is the comparison of change in means for cognitive-behavioral vs. present-centered therapy from baseline to post-treatment for the Perceived Limitations scale; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Net) = -0.47, 95% CI 2-sided [-2.03 to 1.08], Standard Deviation 2.09
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; This is the comparison of change in means for cognitive-behavioral vs. present-centered therapy from baseline to post-treatment for the Satisfaction scale; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Net) = -0.58, 95% CI 2-sided [-2.30 to 1.14], Standard Deviation 2.42

5. Secondary Outcome: Change in Mean Scores on the World Health Organization Disability Assessment Schedule, Version 2.0 (WHO-DAS 2.0) Over 16 Time Points: Baseline, 12 Treatment Sessions, Post-treatment, 3-month and 6-month Follow-up.
Description: The 12-item, self-report version of the WHO-DAS 2.0 will be administered to assess the impact of anger and aggression on broad functioning, as well as across six ICF functioning domains of mobility, self-care, getting along, life activities (household and work) and participation. In addition to the outcome time frame listed above, the WHO-DAS 2.0 will be administered weekly to collect exploratory information about Veterans' perceptions of how their overall functioning changes over the course of the group. The scale range is 0 to 48, with higher scores reflecting greater impairment.
Time Frame: as for outcome 1
Population: For participants without baseline data, the data from the first (of 12) intervention sessions was used as baseline. Last observation carried forward was used for all analyses. Data screening found one participant's data (male, CBT arm) were not valid; his data was not used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 19.3 (8.3) | 24.6 (7.3)
  Post-treatment | 21.6 (9.0) | 20.7 (9.7)
  3 month follow-up | 20.1 (9.4) | 22.4 (8.2)
  6 month follow-up | 22.0 (8.7) | 22.3 (7.7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Estimation parameter is interaction of session by therapy, or estimate of difference in mean between CBT and PCT per time point. Positive value is less decrease over time in CBT arm (greater decrease in anger over time in PCT); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 0.28, Standard Error of Mean 0.06 — The estimation parameter of 0.28 indicates that at each of the 16 time points, participants in the CBT arm had 0.28 point less of a decrease in disability than those in PCT arm

6. Secondary Outcome: Change in Mean Scores on the Inventory of Psychosocial Functioning (IPF) From Baseline to Post-treatment, 3 Month and 6 Month Follow-up.
Description: The IPF is an 80-item self-report measure that assesses functioning over the past 30 days in the following domains: romantic relationships; family relationships; work; friendships and socializing; parenting; academic pursuits; and self-care. The IPF Total score will be used in these analyses. Scores range from 11 to 80, with higher scores reflecting greater functional impairment.
Time Frame: as for outcome 1
Population: Last observation carried forward analyses used; 36 participants assigned to groups. Data screening found one participant's data (male, CBT arm) were not valid; 35 participants' data analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 47.7 (10.7) | 53.4 (15.4)
  Post-treatment | 48.5 (12.7) | 52.7 (14.9)
  3 month follow-up | 50.5 (13.2) | 54.8 (14.1)
  6 month follow-up | 49.2 (10.7) | 55.8 (14.7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Net) = 1.45, Standard Error of Mean 2.71 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Net) = 1.37, Standard Error of Mean 2.71 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Net) = -0.89, Standard Error of Mean 2.71 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

7. Secondary Outcome: The McMaster Family Assessment Device (FAD)
Description: The FAD is a 60-item scale that consists of statements about families to which respondents indicated agreement or disagreement on a 4-point scale. It yields a General Functioning (GF) score, as well as indices of 6 areas of family activity: problem solving; communication; roles; affective responses; affective involvement; and behavioral control. The General Functioning Scale will be used for this outcome. The General Functional Scale scores range from 1-4, with higher scores reflect greater impairment.
Time Frame: pre-treatment, post-treatment, 3 months post-treatment, 6-months post-treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 2.81 (0.61) | 2.50 (0.44)
  Post-treatment | 2.72 (0.49) | 2.60 (0.51)
  3 month follow-up | 2.89 (0.52) | 2.58 (0.51)
  6 month follow-up | 2.86 (0.48) | 2.49 (0.65)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = -0.19, Standard Error of Mean 0.16 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.97, Mixed Models Analysis; Mean Difference (Net) = 0.006, Standard Error of Mean 0.16 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.17 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

8. Other Pre Specified Outcome: The Adaptability Scale of the Connor-Davidson Resilience Scale (CD-RISC)
Description: The Adaptability Scale is an 8-item subscale of the CD-RISC that measures adaptability in the face of challenges (e.g., "I am able to adapt when changes occur"). Cronbach's alpha for the 8-item Adaptability scale was found to be .91 in a sample of 1981Veterans (Green et al, under review). One of the primary goals of the CBT-A intervention is to increase Veterans' behavioral repertoire and range of Activities by targeting maladaptive Thought Functions and Emotion Functions. The Adaptability scale of the CD-RISC will be included among the outcome measures as it may assess improvements in Thought Functions and Emotion Functions that underlie limitations to Activities and Participation. The Adaptability scale scores can range from 0 to 32, with higher scores reflecting better functioning.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 13.4 (3.78) | 13.1 (3.05)
  Post-treatment | 13.5 (3.54) | 13.8 (3.54)
  3 month follow-up | 13.2 (3.37) | 13.4 (3.52)
  6 month follow-up | 12.4 (3.18) | 13.1 (3.54)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = -0.71, Standard Error of Mean 0.66 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.44, Mixed Models Analysis; Mean Difference (Net) = -0.52, Standard Error of Mean 0.66 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -1.06, Standard Error of Mean 0.66 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

9. Other Pre Specified Outcome: PTSD Checklist (PCL)
Description: On the PCL participants first report an autobiographical narrative of a trauma, and subsequently rate symptom frequency (0 [not at all] - 4 [everyday]) and severity (0 [not at all distressing] - 4 [extremely distressing]) for all DSM-V PTSD symptoms within the past week. The PCL will be administered weekly to evaluate the association of PTSD symptoms with anger cognitions (as measured by the DAR) over the course of the group. Total score ranges from 0 to 80, with higher scores reflecting greater impairment.
Time Frame: pre-treatment (baseline), post-treatment (12 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 58.8 (13.2) | 56.0 (12.1)
  Post-treatment | 56.3 (16.4) | 50.8 (17.5)
  3 month follow-up | 57.2 (16.2) | 52.9 (17.7)
  6 month follow-up | 56.1 (15.1) | 52.9 (16.5)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Multilevel model of therapy type (1=CBT, 2=PCT), gender, and time on PCL Total scores, using data from baseline, 12 sessions, post-treatment, 3-month and 6-month follow up; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 0.17, Standard Error of Mean 0.12 — Estimation parameter is interaction of session by therapy, or estimate of difference in mean between CBT and PCT per time point. Positive value is less decrease over time in CBT arm (greater decrease in PTSD in PCT)

10. Other Pre Specified Outcome: The Alcohol Use Disorder Identification Test (AUDIT)
Description: The AUDIT contains 10 multiple choice questions about behavior and symptoms related to alcohol consumption. Scale scores range from 0 to 40, with higher scores reflecting greater impairment. Scores over 8 reflect a strong likelihood of hazardous our harmful alcohol consumption.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 1.89 (2.45) | 3.0 (4.46)
  Post-treatment | 2.11 (2.42) | 2.94 (4.23)
  3 month follow-up | 1.72 (2.11) | 3.06 (4.25)
  6 month follow-up | 1.83 (2.33) | 2.88 (4.03)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = 0.28, Standard Error of Mean 0.37 — Baseline to post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.55, Mixed Models Analysis; Mean Difference (Net) = -0.23, Standard Error of Mean 0.37 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.87, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.37 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

11. Other Pre Specified Outcome: The Drug Abuse Screening Test (DAST)
Description: The DAST contains 20 "yes/no" questions about behavior and symptoms pertaining to substance use. Scale range is 0-20, with higher scores reflecting greater impairment.
Time Frame: pre-treatment (baseline), post-treatment (12 weeks), 3 months post-treatment (48 weeks)
Population: Last observation carried forward analyses used; 36 participants assigned to groups. Data screening found one participant's data (male, CBT arm) were not valid; 35 participants' data analyzed. For one participant (female, PCT), data was available only for 6 month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline: number analyzed (Participants) | 18 | 16
  Baseline | 2.46 (4.24) | 1.27 (1.88)
  Post-treatment: number analyzed (Participants) | 18 | 16
  Post-treatment | 2.11 (3.72) | 1.64 (2.19)
  3 month follow-up: number analyzed (Participants) | 18 | 16
  3 month follow-up | 2.30 (3.74) | 1.52 (1.79)
  6 month follow-up | 2.24 (3.69) | 1.80 (2.15)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = -0.71, Standard Error of Mean 1.04 — Baseline to post-treatment
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Net) = -0.41, Standard Error of Mean 1.04 — Baseline to 3 months post-treatment. The reference condition is the present centered therapy arm
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy vs Present Centered Therapy; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = -0.78, Standard Error of Mean 1.04 — Baseline to 6 months post-treatment. The reference condition is the present centered therapy arm

ADVERSE EVENTS:
Time Frame: AE data were collected from baseline to the 6-month posttreatment visit, which is about 10 months.
Arm/Group | Cognitive Behavioral Therapy | Present Centered Therapy
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=19) | Present Centered Therapy (N=17)
Diagnosed with cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant was diagnosed with stage 4 lung cancer, unrelated to study participation
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pt. was hospitalized due to a collapsed lung, not related to study participation.
Hospitalization (Eye disorders) | 1 (1) | 0 (0) — Pt. was hospitalized after a botched eye surgery, not related to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT02233517/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02233517/ICF_001.pdf